CLINICAL TRIAL: NCT02026492
Title: Exercise-induced Bronchoconstriction in a Cold Chamber Compared to Methacholine Challenge
Brief Title: Exercise Challenge in a Cold Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Consultant Pediatric Allergy and Pneumology, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KGU-208/13
Record Dates: First submitted 2013-12-19; First posted 2014-01-03 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Exercise-induced Asthma
Keywords: exercise-induced bronchoconstriction; exercise-induced asthma; cold chamber; exercise challenge; cold air challenge; combined exercise- and cold-air challenge; methacholine challenge
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 patients aged 6-18 years (Other): All 40 patients with a diagnosis of asthma are recruited from the outpatients clinic of the department of Pediatric Pneumology and Allergology of the University Hospital Frankfurt. Patients undergo a methacholine challenge and two exercise challenges in a cold chamber and one exercise challenge in room temperature.
  Interventions: Other: Exercise challenge in a cold chamber; Other: Methacholine challenge; Other: Exercise challenge in room temperature
- 40 subjects aged 18-45 years (Other): All subjects show bronchial hyperresponsiveness e.g. dyspnea when exercising in cold environment, in their medical history. Subjects undergo a methacholine challenge and exercise challenge in a cold chamber and one exercise challenge in room temperature.
  Interventions: Other: Exercise challenge in a cold chamber; Other: Methacholine challenge; Other: Exercise challenge in room temperature

INTERVENTIONS:
Other: Exercise challenge in a cold chamber — Exercise challenge is defined as running on a treadmill for 6-8 minutes on submaximal work load in a cold chamber.
Other: Methacholine challenge — nebulized metacholine administered at following doses: 0,01mg, 0,1mg, 0,4mg, 0,8mg und 1,6mg
Other: Exercise challenge in room temperature — Exercise challenge is defined as running on a treadmill for 6-8 minutes on submaximal work load in room temperature.

SUMMARY:
The purpose of this study is to compare the exercise-challenge in a cold chamber at 2-4°C to the gold standard the metacholine challenge in subjects showing symptoms of exercise-induced bronchoconstriction. The sensitivity and repeatability of the exercise test will be measured.

DETAILED DESCRIPTION:
Subjects suffering form exercise-induced bronchoconstriction (EIB) usually have a normal lung function testing at rest. To provoke asthma symptoms a provocation test is necessary, e.g., by bronchial methacholine testing or by a standardised exercise test on a treadmill. The correlation between methacholine and exercise test is fair, possibly because both methods measure different kinds of bronchial hyperresponsiveness. Moreover, the sensitivity and the repeatability of the exercise test is fair.

The value of the methacholine test to predict a positive exercise test will be measured. We hypothesize that the exercise test in a cold chamber, a combination of two provocation methods cold air and exercise, is more sensitive to detect EIB and that the test has a better repeatability.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients: Age >6 and <18 years
* Subjects: Age >/=18 and <45 years
* sportive, 1-2x exercise per week
* bronchial hyperresponsiveness in the medical history

Exclusion Criteria:

* lung function Forced vital capacity (FVC) <80% and Forced expiratory volume in 1 second (FEV1) <75%
* chronic diseases or infections (e.g. HIV, Tbc)
* pregnancy
* systemic corticosteroid-treatment
* inhalative corticosteroid therapy or leukotriene antagonists <14d
* alcohol, substance or drug abuse
* smokers
* inability to capture extend and consequences of the study

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Agreement of metacholine challenge and the combined exercise/cold-air challenge | 3 months
  Lung function will be measured prior and after methacholine- and exercise/cold-air challenges. The maximal fall in forced expiratory volume in one second (FEV1, percent predicted) after methacholine and cold air challenge will be compared by statistical correlation. For both methods the sensitivity and the specificity to predict an exercise induced asthma will be calculated by a receiver operating characteristic (ROC analysis).
  All subjects receive Salbutamol to relief them from bronchial constriction at the end of the test.

SECONDARY OUTCOMES:
Repeatability of the combined exercise/cold-air challenge | 3 months
  The combined exercise/cold-air challenge will be performed twice within one week. Post challenge the FEV1 will be measured after 5, 10, 20, and 30 minutes. The maximal fall in FEV1 (percent predicted) and the area under the curve (AUC) will be compared. The agreement and the repeatability of the maximal fall in FEV1 and of the AUC will be measured by correlation and by the method of Bland and Altman.

OTHER OUTCOMES:
Agreement of the combined exercise/cold-air challenge with the Asthma-score | 3 months
  All children who participate will fill the asthma control test (ACT) and all adult subjects will fill the asthma control questionnaire (ACQ). The asthma-score will be compared with the severity of the exercise induced asthma measured by the maximal fall in FEV1.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schulze, MD, Study Chair — Johann Wolfgang Goethe University Hospital
Locations (1):
- Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Schulze J, Rosewich M, Riemer C, Dressler M, Rose MA, Zielen S. Methacholine challenge--comparison of an ATS protocol to a new rapid single concentration technique. Respir Med. 2009 Dec;103(12):1898-903. doi: 10.1016/j.rmed.2009.06.007. Epub 2009 Jul 10. PMID 19596563
- [Background] Anderson SD. Indirect challenge tests: Airway hyperresponsiveness in asthma: its measurement and clinical significance. Chest. 2010 Aug;138(2 Suppl):25S-30S. doi: 10.1378/chest.10-0116. PMID 20668015
- [Background] Parsons JP, Hallstrand TS, Mastronarde JG, Kaminsky DA, Rundell KW, Hull JH, Storms WW, Weiler JM, Cheek FM, Wilson KC, Anderson SD; American Thoracic Society Subcommittee on Exercise-induced Bronchoconstriction. An official American Thoracic Society clinical practice guideline: exercise-induced bronchoconstriction. Am J Respir Crit Care Med. 2013 May 1;187(9):1016-27. doi: 10.1164/rccm.201303-0437ST. PMID 23634861
- [Background] Anderson SD, Charlton B, Weiler JM, Nichols S, Spector SL, Pearlman DS; A305 Study Group. Comparison of mannitol and methacholine to predict exercise-induced bronchoconstriction and a clinical diagnosis of asthma. Respir Res. 2009 Jan 23;10(1):4. doi: 10.1186/1465-9921-10-4. PMID 19161635
- [Background] Driessen JM, van der Palen J, van Aalderen WM, de Jongh FH, Thio BJ. Inspiratory airflow limitation after exercise challenge in cold air in asthmatic children. Respir Med. 2012 Oct;106(10):1362-8. doi: 10.1016/j.rmed.2012.06.017. Epub 2012 Jul 11. PMID 22789953
- [Derived] Dressler M, Friedrich T, Lasowski N, Herrmann E, Zielen S, Schulze J. Predictors and reproducibility of exercise-induced bronchoconstriction in cold air. BMC Pulm Med. 2019 May 16;19(1):94. doi: 10.1186/s12890-019-0845-3. PMID 31097027